CLINICAL TRIAL: NCT07162818
Title: Effects of 0.1% Nepafenac on Vitreous Inflammatory Biomarkers in Rhegmatogenous Retinal Detachment and Proliferative Vitreoretinopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr.dr. Ari Djatikusumo, Sp. M(K)., Head of Ophthalmology Department, Faculty of Medicine Universitas Indonesia Cipto Mangunkusumo Hospital, Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21-01-0081; PUTI Saintekes 2022 Grant (Other: Directorate of Research and Development, Universitas Indonesia)
Record Dates: First submitted 2025-08-25; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Proliferative Vitreoretinopathy; Rhegmatogenous Retinal Detachment
Keywords: Vitreous Inflammatory Biomarker; Nepafenac 0.1%; Proliferative Vitreoretinopathy; Rhegmatogenous Retinal Detachment
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — nepafenac; Ophthalmic Solutions; Population Groups

STUDY DESIGN:
Intervention Model Description: This study will compare the levels of vitreous inflammatory biomarkers in rhegmatogenous retinal detachment (RRD) with proliferative vitreoretinopathy (PVR), following the administration of pre-vitrectomy nepafenac 0.1%, as a method to prevent the progression of PVR.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, the ophthalmologist conducting the eye examinations, and the outcome assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nepafenac 0.1% eyedrops (Experimental): Nepafenac 0.1% is a topical NSAID pro-drug for the eye.
  Interventions: Drug: Nepafenac 0.1% eyedrops
- Control (Placebo Comparator): Cenfresh® sterile eye drops in 5 mL packaging containing 5mg Carmellose sodium
  Interventions: Drug: Control (placebo) group

INTERVENTIONS:
Drug: Nepafenac 0.1% eyedrops — The study eye drops were nepavenac 0.1% eye drops (NEVANAC 0.1%®, Alcon Laboratories, Inc., Fort Worth, Texas). Subjects were instructed to use eye drops on the side of the eye with the ARR, three times daily for five days before and on the day of surgery. Written instructions and a daily checklist to record the eye drop schedule were provided to each subject.
  Arms: Nepafenac 0.1% eyedrops
Drug: Control (placebo) group — Cenfresh® eye drops (Cendo pharmaceutical, Indonesia) for the control group. Subjects were instructed to use eye drops on the side of the eye with the ARR, three times daily for five days before and on the day of surgery. Written instructions and a daily checklist to record the eye drop schedule were provided to each subject.
  Arms: Control

SUMMARY:
PVR remains the major cause of surgical failure in RRD repair.1 Prompt surgical management is the standard therapy in RRD repair. However, in many places, vitreoretinal (VR) surgery facilities is limited, such as in Indonesia, where mainly located within referral hospitals. Until recently, there has been no recommended pharmacological therapy before surgery to prevent the formation of PVR in RRD. . Previous studies involving the use of pharmacological agents, such as anti-inflammatory and anti-proliferative agents, have been reported to prevent the development of PVR. Nepafenac 0.1% eye drops is a potent NSAID that has been proven effective in preventing macular edema in cases of post-cataract surgery and diabetic retinopathy. This study aims to compare the levels of vitreous inflammatory biomarkers in RRD following the administration of preoperative nepafenac 0.1%.

The inclusion criteria were patients of the age of 18 years old and above with macula-off RRD, grade A or B PVR, and RRD onset upon examination up to 1 month. The exclusion criteria included RRD patients with media opacification, a history of intraocular surgery in less than 3 months, other eye disease comorbidities (i.e., macular hole, epiretinal membrane), other systemic diseases, and a history of NSAID allergy.

DETAILED DESCRIPTION:
Prospective subjects underwent Vital signs, an eye examination, fundus biomicroscopy, fundus photographs, and an Optical Coherent Tomography (OCT) scan of the macula were performed. This initial eye examination determined the degree of PVR before intervention was administered.

If they met the inclusion criteria, potential subjects were recruited and randomized, allocating the subjects to two groups: an intervention group with nepavenac 0.1% eye drops and a control group with Cenfresh® eye drops, administered 5 days before the vitrectomy. The medication labels were removed and replaced with the study labels.

The subjects were then prepared for surgery by undergoing blood tests, an EKG, and consultation with an anesthesiologist in the perioperative clinic of the Department of Anesthesia, RSCM/FKUI. The surgery was performed in the operating room of the Department of Ophthalmology, FKUI/RSCM Kirana, according to a predetermined schedule, which was after the subjects had used the eye drops for 5 days, 3 times daily. Written instructions and a daily checklist to record the medication drop schedule were provided to each subject.

On the day of surgery, a repeat fundus biomicroscopy examination, fundus photographs, and an OCT macular scan were performed to record the degree of PVR before the vitrectomy. Vitreous samples were taken during vitrectomy to assess vitreous biomarker levels.

After vitrectomy, all subjects underwent follow-up examinations on days 1, 7, and 28 to assess the surgical outcome. At each visit, routine examinations were performed, including vital signs, an eye examination, and fundus biomicroscopy. Fundus photographs and OCT scans were performed three times:

On the first visit during recruitment, the second visit on the day of surgery, and the final one on day 28 postoperatively. All examination results were recorded in the outpatient record at each visit.

ELIGIBILITY:
Inclusion Criteria:

* ARR with PVR grade A and B
* ARR onset more than 7 days and less than 1 month
* Macula off
* ARR patients with a minimum age of 18 years.
* Willing to follow the research stages and sign the informed consent.

Exclusion Criteria:

* ARR patients with media opacities that do not allow fundus examination
* History of undergoing intraocular surgery less than 3 months.
* ARR patients with comorbid eye diseases.
* ARR patients with systemic complications that make it impossible to undergo vitrectomy surgery.
* ARR sufferers who are known to have a history of allergies to the NSAID group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Prostaglandin E2 (PGE2) | Through study completion, an average of 1 year
  Vitreous samples were thawed and prostaglandin E2 (PGE2) levels were analyzed using the Prostaglandin E2 Monoclonal ELISA Kit (Cayman Chemical Company, Ann Arbor, MI) using a competitive ELISA according to the manufacturer's instructions. Briefly, serial dilutions of standards (7.8-1000 pg/mL) were prepared. Standards, controls, and vitreous samples were added to microplate wells coated with a specific polyclonal antibody against mouse IgG, followed by the addition of the acetylcholinesterase-PGE2 conjugate tracer and the PGE2 monoclonal antibody. The plates were incubated overnight at 40°C. During incubation, competition occurred between PGE-2 in the samples/standards and the PGE2 monoclonal antibody. The PGE-2 antibody complex bound to the polyclonal antibody against mouse IgG on the well walls. The plate was washed, then Ellman's reagent was added to each well of the microplate. The plate was covered and incubated at room temperature on an orbital shaker for 60 minutes. The color f
Transforming Growth Factor β1 (TGF-β1) | Through study completion, an average of 1 year
  Vitreous samples were thawed and activated before the sandwich ELISA test using the Quantikine ELISA Human TGFβ-1 kit (R&D Systems, MN, USA). Activation was performed by placing 40 μL of sample in a tube and adding 20 μL of 1N HCl, which was incubated for 10 minutes at room temperature. Next, the sample was neutralized by adding 20 μL of 1.2N NaOH and 0.5 M HEPES. Afterward, the sample was diluted 1:20 with RD5-53 calipers (a 1:4 dilution). Fifty μL of RD1-73 solution was added to each well of the microplate, followed by 50 μL of sample or standard, and incubated for 2 hours at room temperature. After the incubation period, the plate was washed three times with 400 μL of buffer. Afterward, anti-TGFb-1 conjugate was added to each well and incubated for another 2 hours at room temperature. After incubation, a wash was performed, then 100 μL of substrate solution was added, incubated for another 13 minutes at room temperature, protected from light, and the reaction was stopped by adding
Siklooksigenisase-2 (COX-2) Enzyme | Through study completion, an average of 1 year
  Vitreous samples were thawed and activated before the sandwich ELISA assay using the Human Cyclooxygenase 2 (COX-2) kit according to the protocol. The vitreous samples were added to the wells of a microtiter plate coated with a monoclonal antibody against COX-2. If COX-2 is present in the sample, it will bind to the antibody. To quantitatively determine the amount of COX-2 in the sample, standards with varying concentrations of COX-2 were added. After incubation, the COX-2 antibody on the well walls binds to the COX-2 in the sample or standard. After washing to remove any unbound components, a horseradish peroxidase (HRP)-conjugated polyclonal antibody was added. The microtiter plate was incubated and then washed. Next, substrate solution was added to each well of the microtiter plate. The HRP enzyme and substrate were allowed to react for a short incubation period. Only wells containing COX-2 showed a color change due to binding to the HRP-conjugated antibody. The enzyme-substrate re
Macrophage Cell Count | Through study completion, an average of 1 year
  The number of macrophages in vitreous samples was measured using flow cytometry, utilizing CD14 as a monocyte/macrophage marker. Pure vitreous samples were prepared according to a modification of the protocol adopted for cytology samples at the Faculty of Medicine, University of Indonesia (FKUI) Integrated Laboratory. After incubation for 10 minutes at room temperature in the dark, the samples were centrifuged for 5 minutes at 1500 rpm. The supernatant was discarded and washed with 2.5 mL of buffer solution. Antibody was added, and the samples were then incubated in the dark at room temperature for 20 minutes. After 20 minutes, excess antibody was washed away with buffer solution. Flow cytometry was performed using a FACSCanto II flow cytometer (Becton Dickinson, San Jose, CA). The results were analyzed using the FACSDiva program.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Djatikusumo, MD, Principal Investigator — Department of Ophthalmology, Faculty of Medicine Universitas Indonesia Cipto Mangunkusumo Hospital, Indonesia
Locations (1):
- Department of Ophthalmology, Faculty of Medicine Universitas Indonesia Cipto Mangunkusumo Hospital, Jakarta, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No